CLINICAL TRIAL: NCT05428098
Title: The Effect of educatıon and counselıng gıven to patıents patıent wıth Prostatectomy on qualıty of lıfe
Brief Title: The Effect of the Educatıon and Counselıng of Prostatectomy Patıents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Sevgi Deniz Dogan, lecturer Dr., Cukurova University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 5312256941
Record Dates: First submitted 2022-06-15; First posted 2022-06-22 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer; Surgery; Nursing Caries
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (Experimental): In addition to standard care, patients will be given discharge training, planned within the framework of the Life model, one day before discharge. It is planned that the discharge training will be given by the researcher in the patient's room and by providing an accompanying person. Written training material will be delivered to the patients for their re-use after the training.
  Interventions: Other: education
- control group (No Intervention): standard care will be applied

INTERVENTIONS:
Other: education — Oral and written education according to the life model
  Arms: experiment group

SUMMARY:
The research was planned as a randomized controlled experimental study. This study is planned to be conducted in the Urology clinic of a university hospital located in the south of Turkey. The population of the research will be the patients admitted to the urology clinic for prostatectomy. The sample of the study will consist of patients who meet the criteria for participation in the study and volunteer to participate in the study. Evaluation of the research data will be done with the SPSS package program.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* Being literate,
* Being able to understand and speak Turkish and not have a hearing impairment,
* Agreeing to participate in the research.

Exclusion Criteria:

* Development of any complications during the surgical intervention,
* Having any psychiatric disorder that will reduce the ability to comprehend and understand,
* Having other concomitant cancer,
* Having metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male patients will be covered due to the surgical procedure.
Enrollment: 42 (Actual)
Dates: Start 2022-07-10 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Effect of traınıng and counselıng gıven after prostatectomy on qualıty of lıfe | six months
  It will be measured with SF-12. Measurement will be made before and after the application. It is evaluated between 0 and 100 points, with a higher score representing better health.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)